CLINICAL TRIAL: NCT00749359
Title: An Open-label, Randomized, Single Dose, Two-period Crossover Study to Demonstrate Bioequivalence Between the Controlled Release Paroxetine Tablet (37.5 mg) Manufactured at Cidra and Mississauga
Brief Title: PAXIL CR Bioequivalence Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: PCR111656
Record Dates: First submitted 2008-09-05; First posted 2008-09-09 (Estimated); Last update posted 2017-08-04 (Actual); Status verified 2017-08

CONDITIONS: Depressive Disorder
Keywords: healthy volunteers; paroxetine
MeSH Terms: conditions — Depressive Disorder | interventions — Paroxetine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- open label treatment (Experimental): On each treatment period, subjects will receive controlled release paroxetine 37.5 milligram (mg) on Day 1.
  Interventions: Drug: Paxil CR

INTERVENTIONS:
Drug: Paxil CR — Paxil CR 37mg tablet manufactures at two different sites

SUMMARY:
This study is to determine if controlled release paroxetine tablets manufactured at two different sites behave similarly in healthy volunteers.

ELIGIBILITY:
Key Inclusion:

Healthy males or females between 18-65. Body weight 50 kg (110 lbs) or higher, and BMI within the range 19-30 kg/m2. Willing to use acceptable forms of birth control throughout the study. Normal labs and ECG.

Key Exclusion:

Positive test for drugs or alcohol. Positive for Hepatitis or HIV. Any history of psychiatric disorder or suicidal behavior. Has taken another investigational product within 30 days of the start of this study. Has been exposed to more than 4 new chemical entities in the last 12 months. Females who are pregnant or nursing. Regular consumption of alcohol; >14 drinks/week for men or >7 drinks/week for women. Heavy smokers; greater than 20 cigarettes per day.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 166 (Actual)
Dates: Start 2008-07-07 (Actual); Primary Completion 2008-09-16 (Actual); Study Completion 2008-09-16 (Actual)

PRIMARY OUTCOMES:
Paroxetine blood levels | measured up to 168 hours after a single dose.

SECONDARY OUTCOMES:
Additional pharmacokinetic parameters related to blood levels of paroxetine . Safety & tolerability measures including ae reporting & vitals signs & ECGs | measured up to 168 hours after a single dose and throughout study

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (2):
- United States (2):
  - GSK Investigational Site, Buffalo, New York
  - GSK Investigational Site, Tacoma, Washington

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- See also: Results for study PCR111656 can be found on the GSK Clinical Study Register. — https://www.gsk-clinicalstudyregister.com/study/PCR111656?search=study&search_terms=PCR111656#rs
- Available data/document: Study Protocol: PCR111656 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: PCR111656 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: PCR111656 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: PCR111656 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: PCR111656 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: PCR111656 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: PCR111656 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register